CLINICAL TRIAL: NCT04503668
Title: Phase III Randomized Control Trial Investigating Olanzapine for the Prevention of Chemotherapy Induced Nausea and Vomiting in Patients With Gynecologic Malignancies Receiving Every 3-week Carboplatin and Paclitaxel Chemotherapy
Brief Title: Olanzapine for the Prevention of Chemotherapy Induced Nausea and Vomiting in Gynecologic Oncology Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of Patient Population
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2019.173; HUM00175458 (Other: University of Michigan)
Record Dates: First submitted 2020-08-03; First posted 2020-08-07 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Gynecologic Cancer
MeSH Terms: interventions — Ondansetron; Dexamethasone; Neurokinin-1 Receptor Antagonists; fosaprepitant; Olanzapine; Prochlorperazine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nk1-RA (Active Comparator): Nk1-RA will be given on day 1 of each 3-week chemotherapy cycle, for up to 6 cycles.
  Interventions: Drug: Ondansetron; Drug: Dexamethasone; Drug: Neurokinin-1 Receptor Antagonist (NK1-RA); Drug: Compazine
- Olanzapine (Experimental): Olanzapine will be given on days 1-4 of each 3-week chemotherapy cycle, for up to 6 cycles.
  Interventions: Drug: Ondansetron; Drug: Dexamethasone; Drug: Olanzapine; Drug: Compazine

INTERVENTIONS:
Drug: Ondansetron — 8 mg IV or 16 mg by mouth on day 1 pre-chemotherapy; then 8 mg by mouth twice a day on days 2-4 of chemotherapy
Drug: Dexamethasone — 20 mg IV on day 1 pre-chemotherapy
Drug: Neurokinin-1 Receptor Antagonist (NK1-RA) — 150 mg IV on day 1 pre-chemotherapy
  Other Names: Fosaprepitant
  Arms: Nk1-RA
Drug: Olanzapine — 5 mg by mouth on days 1-4 of chemotherapy (taken at night)
  Other Names: Zyprexa
  Arms: Olanzapine
Drug: Compazine — 5-10 mg by mouth, available as needed, every 6 hours, days 1-5

SUMMARY:
The objective of this study is to investigate the efficacy of olanzapine as compared to neurokinin-1 receptor antagonists (NK1-RAs) in the prevention of chemotherapy-induced nausea and vomiting (CINV) in patients with gynecologic malignancies receiving single day outpatient chemotherapy (carboplatin and paclitaxel) every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gynecologic malignancy
* No chemotherapy in the last 12 months
* Scheduled to receive Carboplatin (AUC>=4) and Paclitaxel every three weeks
* ECOG performance status 0 or 1
* English speaking
* Willing and able to provide informed consent
* Laboratory values within protocol-defined parameters
* No vomiting in the 24 hours prior to initiating chemotherapy
* If childbearing potential exists, negative pregnancy test within 7 days prior to registration

Exclusion Criteria:

* Significant cognitive compromise
* History of CNS disease (e.g. brain metastases, seizure disorder, dementia)
* Current or recent (within 30 days) treatment with another antipsychotic agent (antidepressant medications are OK)
* Concurrent radiotherapy treatment
* Known hypersensitivity to olanzapine
* Known cardiac arrhythmia, uncontrolled congestive heart failure or acute myocardial infarction within the last six months
* History of diabetes mellitus on medication (insulin or oral glycemic agent)
* Alcohol abuse / chronic alcoholism
* History of closed angle glaucoma
* Current enrollment in other clinical trials

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Rolston, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nk1-RA | Olanzapine
Started | 31 | 31
Completed | 24 | 27
Not Completed | 7 | 4
Not completed — Incomplete data | 4 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nk1-RA | Olanzapine | Total
Number analyzed (Participants) | 27 | 24 | 51
Age, Customized [Mean (Full Range); unit: years]
  Age | 69 [64 to 73] | 72 [61 to 74] | 69 [61 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 25 | 23 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 27 | 24 | 51

OUTCOME MEASURES:

1. Primary Outcome: Rate of Complete Response in the Overall Time Period (0 - 120 Hours Post-chemotherapy)
Description: Complete response (CR) is defined as no episodes of vomiting and no use of rescue antiemetic medications. Patient reported diaries will be used to measure this outcome.
Time Frame: 120 hours post initiating chemotherapy during cycle 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nk1-RA | Olanzapine
Number analyzed (Participants) | 27 | 24
Participants | 11 | 14

2. Secondary Outcome: Rate of Complete Response in the Acute Time Period (0 - 24 Hours Post-chemotherapy)
Description: as for outcome 1
Time Frame: 24 hours post initiating chemotherapy during cycle 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nk1-RA | Olanzapine
Number analyzed (Participants) | 27 | 24
Participants | 19 | 22

3. Secondary Outcome: Rate of Complete Response in the Delayed Time Period (24 - 120 Hours Post-chemotherapy)
Description: as for outcome 1
Time Frame: 24-120 hours post initiating chemotherapy during cycle 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nk1-RA | Olanzapine
Number analyzed (Participants) | 27 | 24
Participants | 14 | 14

4. Secondary Outcome: Rate of no Nausea in the Acute Time Period (0 - 24 Hours Post-chemotherapy)
Description: Patients will record daily levels of nausea after chemotherapy using a Likert scale ranging from 0-10 (0 indicating no nausea; 10 indicating maximum level of nausea).
Time Frame: 24 hours post initiating chemotherapy during cycle 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nk1-RA | Olanzapine
Number analyzed (Participants) | 27 | 24
Participants | 17 | 19

5. Secondary Outcome: Rate of no Nausea in the Delayed Time Period (24 - 120 Hours Post-chemotherapy)
Description: Patients will record daily levels of nausea using a Likert scale ranging from 0-10 (0 indicating no nausea; 10 indicating maximum level of nausea).
Time Frame: 120 hours post initiating chemotherapy during cycle 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nk1-RA | Olanzapine
Number analyzed (Participants) | 27 | 24
Participants | 10 | 8

6. Secondary Outcome: Rate of no Nausea in the Overall Time Period (0 - 120 Hours Post-chemotherapy)
Description: as for outcome 5
Time Frame: 120 hours post initiating chemotherapy during cycle 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nk1-RA | Olanzapine
Number analyzed (Participants) | 27 | 24
Participants | 9 | 6

7. Secondary Outcome: Mean Somnolence Score
Description: Patients will record daily levels of undesired sedation using a Likert scale ranging from 0 to 10 (0 indicating no undesired sedation; 10 indicating maximum level of undesired sedation).
Time Frame: assessed daily, and reported at day 6 post final study treatment
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Nk1-RA | Olanzapine
Number analyzed (Participants) | 27 | 24
score on a scale | 0.81 [0.13 to 1.49] | 1.15 [0.39 to 1.93]

8. Secondary Outcome: Mean Increased-appetite Score
Description: Patients will record daily levels of undesired increase in appetite using a Likert scale ranging from 0 to 10 (0 indicating no undesired increase in appetite; 10 indicating maximum level of undesired increase in appetite).
Time Frame: assessed daily, and reported at day 6 post final study treatment
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Nk1-RA | Olanzapine
Number analyzed (Participants) | 27 | 24
score on a scale | 0.45 [0.06 to 0.85] | 0.33 [0.09 to 0.56]

ADVERSE EVENTS:
Time Frame: All adverse event data (serious and non-serious) collected from the time of the initial study treatment administration through 30 days after the last dose of study treatment. Up to 2 years. Adverse Events will be evaluated with secondary endpoints
Description: Adverse Events and All-Cause Mortality will be evaluated with secondary endpoints
Arm/Group | Nk1-RA | Olanzapine
All-Cause Mortality (participants affected / at risk) | 4/27 | 6/24
Serious Adverse Events (participants affected / at risk) | 3/27 | 5/24
Other Adverse Events (participants affected / at risk) | 24/27 | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nk1-RA (N=27) | Olanzapine (N=24)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
anemia (Investigations) | 1 (1) | 0 (0)
syncope (Nervous system disorders) | 1 (1) | 0 (0)
fall (General disorders) | 1 (1) | 0 (0)
dizziness (General disorders) | 1 (1) | 0 (0)
hyponatremia (Investigations) | 1 (1) | 0 (0)
creatinine increased (Investigations) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
debulking surgery (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nk1-RA (N=27) | Olanzapine (N=24)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 8 (9) | 8 (10)
abdominal cramping (Gastrointestinal disorders) | 2 (2) | 0 (0)
abdominal distention (Gastrointestinal disorders) | 2 (2) | 1 (1)
alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1)
alkaline phosphatase increased (Investigations) | 5 (5) | 2 (3)
alopecia (General disorders) | 6 (7) | 2 (2)
anemia (Investigations) | 10 (18) | 6 (8)
anorexia (Psychiatric disorders) | 1 (1) | 3 (3)
arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 6 (10)
aspartate aminotransferase increased (Investigations) | 2 (2) | 3 (3)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
bloating (Gastrointestinal disorders) | 2 (2) | 1 (1)
cognitive disturbance (General disorders) | 2 (2) | 0 (0)
constipation (Gastrointestinal disorders) | 7 (7) | 10 (14)
creatinine increased (Investigations) | 2 (2) | 2 (3)
diarrhea (Gastrointestinal disorders) | 3 (5) | 9 (10)
dizziness (General disorders) | 5 (6) | 0 (0)
dry mouth (General disorders) | 2 (2) | 0 (0)
dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2)
edema limbs (General disorders) | 1 (1) | 2 (2)
facial flushing (General disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 19 (27) | 11 (12)
headache (General disorders) | 4 (6) | 4 (4)
hypoalbuminemia (Investigations) | 2 (2) | 0 (0)
hypocalcemia (Investigations) | 2 (2) | 2 (4)
hypokalemia (Investigations) | 3 (3) | 2 (2)
hypomagnesemia (Investigations) | 2 (2) | 0 (0)
hyponatremia (Investigations) | 3 (3) | 4 (4)
Insomnia (Psychiatric disorders) | 4 (4) | 2 (3)
lymphocyte count decreased (Investigations) | 6 (8) | 2 (3)
myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 6 (8)
nausea (Gastrointestinal disorders) | 12 (19) | 15 (20)
neuropathy (Nervous system disorders) | 4 (5) | 5 (5)
neutropenia (Investigations) | 0 (0) | 2 (2)
peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 5 (6)
platelet count decreased (Investigations) | 5 (7) | 2 (4)
presyncope (Cardiac disorders) | 2 (2) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
vomiting (Gastrointestinal disorders) | 1 (2) | 6 (9)
white blood cell decreased (Investigations) | 2 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/68/NCT04503668/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/68/NCT04503668/ICF_001.pdf